CLINICAL TRIAL: NCT03314961
Title: Localisation of Mesenteric Lymph Node Metastases and Role of Level of Arterial Ligation in Rectal Cancer Surgery
Brief Title: Lymph Node Metastases and Arterial Ligation in Rectal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Catarina Tiselius, MD, PhD, Region Västmanland
Other Study IDs: Dnr2013/099
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Lymph Node Metastases
Keywords: rectal cancer
MeSH Terms: conditions — Lymphatic Metastasis; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lymph node status is of major prognostic importance in non-metastatic rectal cancer. For oncological reasons, central arterial ligation of the inferior mesenteric artery (IMA) is suggested. However, there is no conclusive evidence presented for this procedure.

This study aimed at investigating the localisation of lymph node metastases and the role of central versus peripheral arterial ligation of in rectal cancer specimens.

DETAILED DESCRIPTION:
Prospective population-based study of specimens from patients that underwent surgical resection for rectal cancer in Västmanland County, Sweden. Specimens were divided in 3 sections (A-C) and the total amount of lymph nodes and the location of lymph node metastases were analysed.

Multivariate analysis was used to explore the relationship between lymph node counts and age, gender, BMI, preoperative oncological treatment, type of surgery, tumour stage, vessel and specimen length.

ELIGIBILITY:
Inclusion Criteria:

* All patients that were curatively operated for rectal cancer in Västmanlands county 2012-2016.

Exclusion Criteria:

* Patients that were not operated or had another type of cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that were diagnosed with rectal cancer 2012-2016 in Västmanlands county.
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Lymph node metastases in rectal cancer | 2012-2016
  Analyses of number and location of lymph node metastases in rectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Tiselius, MD, PhD, Principal Investigator — Region Västmanland

IPD SHARING:
Plan to Share IPD: No